CLINICAL TRIAL: NCT02249390
Title: ART Survey: Assisted Reproductive Technology Survey
Brief Title: Assisted Reproductive Technology Survey (ART Survey)
Acronym: ART
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Leanne Redman, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 2014-042
Record Dates: First submitted 2014-09-18; First posted 2014-09-25 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Female Reproductive Problem; Male Reproductive Problem

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anyone: Any individual may complete this survey

SUMMARY:
The purpose of the study is to collate local information to better understand the motivations, accessibility and frequency of assisted reproductive technology (ART) use in the community.

DETAILED DESCRIPTION:
The ART survey study recruitment will last about 6 months with the study completed within 1 year. Study participation is an online survey which takes approximately 3 minutes to complete.

The goal is to apply for future funding to study the metabolic consequences of being conceived with ART.

ELIGIBILITY:
Inclusion Criteria:

* Any individual may complete this survey

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited from the community. Parents of children who have participated in a research study at Pennington Biomedical Research Center or patients from local fertility clinics.
Sampling Method: Non-Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2014-09; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Method of Conception | 1 year
  ART Survey

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Redman, MS, PHD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States